CLINICAL TRIAL: NCT00656006
Title: A Randomized, Multi-Center, Open-Label Study To Evaluate The Efficacy And Safety Of Albuferon (HGS 1008, Recombinant Human Albumin-Interferon Alfa Fusion Protein) In Combination With Ribavirin In Interferon Alfa Naive Subjects With Chronic Hepatitis C Genotype 2 OR 3
Brief Title: A Study of Albuferon With Ribavirin in Interferon Alfa Naive Subjects With Chronic Hepatitis C Genotype 2 or 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Patrick Cronin, Human Genome Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGS1008-C1052 (ALFR-HC-06)
Record Dates: First submitted 2005-12-20; First posted 2008-04-10 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Chronic; Genotype 2 or 3; Treatment naive
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Bronchiolitis Obliterans Syndrome | interventions — albuferon; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Albuferon
Drug: Ribavirin

SUMMARY:
A Study of Albuferon with Ribavirin in Interferon Alfa Naive Subjects with Chronic Hepatitis C Genotype 2 or 3.

DETAILED DESCRIPTION:
A Randomized, Multi-Center, Open-Label Study To Evaluate The Efficacy And Safety Of Albuferon (HGS 1008, Recombinant Human Albumin-Interferon Alfa Fusion Protein) In Combination With Ribavirin In Interferon Alfa Naive Subjects With Chronic Hepatitis C Genotype 2 OR 3

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of chronic hepatitis C on the basis of detectable serum HCV RNA during the screening period and at least a 6-month history of exposure to risk factors for HCV.
* Have never received treatment with an interferon alfa product or an interferon alfa combination product.
* Have HCV genotype 2 or 3.
* Have compensated liver disease with the following minimum criteria: white blood cell count (WBC) >3,000/mm3, absolute neutrophil count (ANC) > 1,800/mm3, platelets >100,000/mm3, hemoglobin (Hb) > 13 g/dL for males and > 12 g/dL for females.

Exclusion Criteria:

* Evidence of decompensated liver disease.
* Pregnant or lactating female.
* History of any other medical disease or condition that would make the subject (in the opinion of the investigator) unsuitable for the study.
* A current drug or alcohol addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Primary safety endpoints are the common side effects of IFNa therapy including flu-like symptoms, depression, and hematologic abnormalities.
Primary efficacy end point is sustained virologic response (SVR), defined as undetectable HCV RNA at 24 weeks after the end of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - University of Western Ontario, London, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan